CLINICAL TRIAL: NCT05104372
Title: Hypertonic Saline Nasal Irrigation and Gargling (HSNIG) for Suspected COVID-19: Pragmatic, Web-based Bayesian Adaptive Randomised Controlled Trial in Pakistan
Brief Title: Hypertonic Saline Nasal Irrigation and Gargling (HSNIG) for Suspected COVID-19 in Pakistan
Acronym: HSNIG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Allergy and Asthma Institute, Pakistan (Other)
Collaborators: University of Edinburgh (Other)
Responsible Party: Principal Investigator, Osman Yusuf, Chief Consultant, The Allergy and Asthma Institute, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16/136/109-AAIP-NW
Record Dates: First submitted 2021-10-25; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Mouthwashes

STUDY DESIGN:
Intervention Model Description: A randomised intervention and a control arm, running in parallel
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention Group HSNIG started within 5 days of symptom onset Number of times HSNIG should be done: As many times as needed (but not more than 12 times/day) PLUS
  Standard personal, household hygiene and social distancing advice:
  http://www.covid.gov.pk/prevention
  Interventions: Other: Hypertonic Saline Nasal Irrigation and Gargles (HSNIG)
- Control (Placebo Comparator): Control Group
  Standard personal, household hygiene and social distancing advice:
  http://www.covid.gov.pk/prevention
  Interventions: Other: Hypertonic Saline Nasal Irrigation and Gargles (HSNIG)

INTERVENTIONS:
Other: Hypertonic Saline Nasal Irrigation and Gargles (HSNIG) — Nasal washout and gargles

SUMMARY:
Nasal washing (washout) followed by gargles with hypertonic saline (HSNIG) is believed to be effective in reducing the duration of illness in those with clinically suspected or confirmed COVID-19 being managed at home, and also is effective in reducing complications of COVID-19 and onward household transmission.

This study plans to investigate whether the use of HSNIG performed by adults with symptoms consistent with COVID-19 reduces the duration of symptoms when compared to participants managed using standard care.

DETAILED DESCRIPTION:
BACKGROUND

Analysis of data from the recent "Edinburgh and Lothians Viral Intervention Study" (ELVIS) pilot randomized controlled trial (RCT) indicates that hypertonic saline nasal irrigation and gargling (HSNIG) reduced the duration of coronavirus upper respiratory tract infection (URTI) by an average of two-and-a-half days. As such, it may offer a potentially safe, effective and scalable intervention in those with Coronavirus Disease-19 (COVID-19) following infection with the beta-coronavirus Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2).

The researchers recently reported that epithelial cells mount an antiviral effect by producing hypochlorous acid (HOCl) from chloride ions. HOCl is the active ingredient in bleach. Epithelial cells have this innate antiviral immune mechanism to clear viral infections. Since bleach is effective against all virus types, it was tested to see whether a range of DNA, RNA, enveloped and non-enveloped viruses were inhibited in the presence of chloride ions supplied via salt (NaCl). All the viruses tested were inhibited in the presence of NaCl. The human viruses which were tested included: DNA/enveloped: herpes simplex virus; RNA/enveloped: human coronavirus 229E (HCoV-229E), respiratory syncytial virus, influenza A virus; and RNA/non-enveloped: coxsackievirus B3.

In COVID-19, high titers of SARS-CoV-2 are detectable in the upper respiratory tract of asymptomatic and symptomatic individuals. The titers are higher in the nose than the throat suggesting measures that control the infection and viral shedding will help reduce transmission.

Till the time a significant proportion of the world population is vaccinated against COVID-19, a safe and effective intervention is needed that can be implemented globally. The in-vitro data gives the evidence that NaCl has an antiviral effect that works across viral types. The findings from this post-hoc analysis of ELVIS need to be interpreted with caution. These data do however suggest that HSNIG may have a role to play in reducing symptoms and duration of illness in COVID-19.

HYPOTHESES Primary: HSNIG is effective in reducing the duration of illness in those with clinically suspected or confirmed COVID-19 being managed at home.

Secondary: HSNIG is effective in reducing complications of COVID-19 and onward household transmission.

INTERVENTION The Intervention group will be suspected or confirmed COVID-19 infected individuals. They will make hypertonic saline at home, and perform nasal washing and gargles, as per instructions and study videos, which will be available to be viewed by the intervention group only, in the study website "www.nasalwash.pk". This will be used as required to a maximum of 12 times/day for a maximum of 14 days. Participants are informed that symptoms might reduce after HSNIG, but may return after a while. Symptoms could hence return as early as 30 minutes to many hours after HSNIG. Participants will be advised to perform HSNIG as soon as symptoms return, and as many times as needed (but not more than 12 times/day) until they become symptom-free, or until the end of their study participation (either on day 14, or on admission to hospital or on withdrawal from the study), and follow standard advice from their physicians or the Pakistan Government website on personal and household hygiene and social distancing: http://www.covid.gov.pk/prevention.

CONTROL The participants randomized to the control arm will be asked to perform ablution, which includes washing of the nose by the prescribed Islamic method with plain water, (instructions and study videos are available to be viewed by the control group in the study website) and to follow the guidance on personal and household hygiene and social distancing as advised by the Ministry of Health, Government of Pakistan, at http://www.covid.gov.pk/prevention.

OBJECTIVES Primary Objective To investigate whether the use of HSNIG performed by adults with symptoms consistent with COVID-19 reduces the duration of symptoms when compared to participants managed using standard care.

Secondary Objectives

To determine the effect of HSNIG on:

1. Severity of all symptoms
2. Duration and severity of individual symptoms
3. Over-the-counter medication use
4. Contact with primary care, or Covid19 emergency helpline.
5. Hospital emergency attendance and/or hospital admission, and diagnosis
6. Number of household contacts infected
7. Side-effect of HSNIG.

ENDPOINTS Primary Endpoint Self-reported time to resolution as assessed by completion of the validated self-reported UK-adapted short form of the Wisconsin Upper Respiratory Symptom Survey (WURSS-24) which will be used to collect daily symptom data.

Secondary Endpoints

1. Severity of all symptoms
2. The length of time for individual symptoms to resolve
3. Severity of individual symptoms
4. Contacting healthcare.
5. Participants needing physician appointments.
6. Participants attending hospital
7. Length of stay in hospital, if admitted
8. Number of participants reporting over the counter medication use
9. Reduction in transmission to household contacts
10. Number of participants reporting side effects of nasal irrigation
11. Types and severity of side effects reported

STUDY DESIGN

This study is a pragmatic, non-CTIMP, web-based, Bayesian adaptive randomized controlled trial (RCT) of HSNIG vs. standard care in adults over 18 years of age with suspected or confirmed COVID-19. The study will run throughout the course of the COVID-19 pandemic until numbers have been recruited for sufficient analysis, or until 30th of November 2021. Participants are recruited within 5 days of developing COVID-19 symptoms by use of the study website ("www.nasalwash.pk"), study advertising through traditional media such as radio and internet advertisements, as well as social media. Paper leaflets will be distributed at chemists, doctors' clinics, COVID testing centers, and through organizations working with COVID patients. For the purposes of this study, symptoms or diagnosis of COVID-19 are defined as at least one of the following symptoms, which include:

* Respiratory symptoms, such as cough and shortness of breath
* Fever
* Muscle pain
* Headache
* Sore throat
* New loss of taste or smell
* Severe fatigue
* Nausea or vomiting
* Diarrhea
* Congestion or runny nose

Willing participants will be directed by the study advertising to a study specific webpage at "www.nasalwash.pk", where they will be able to access further study information and documents, which will include a Patient Information Sheet and a Consent form. All data including consent will be obtained electronically, details of how the process of electronic consent will work is given in detail below in the section titled "Consenting Participants".

After obtaining their electronic consent, they will be randomized automatically by the software to either the Intervention Group, or the Control Group. They will be provided a password to a personal area, which will contain an instructional video on whether they will perform hypertonic saline nasal irrigation and gargles (the intervention group); or do either nothing, or regularly continue to perform ablution for prayers (the control group). The affected individual (not more than one participant per household) will be centrally randomized through an easy to access web-based randomization schedule hosted at the study data center at the Allergy & Asthma Institute, Pakistan, in collaboration with the Edinburgh Clinical Trials Unit, University of Edinburgh.

All pre- and post-randomization data will be collected through mobile phone/web-based questionnaires (see Daily Study Diary, Daily Symptom report, End of Illness questionnaire and Day 14 questionnaire). Participants will be randomized to either a Control arm of standard symptomatic care, or an Intervention arm of HSNIG up to 12 times per day for a maximum of 14 days or until asymptomatic, alongside standard symptomatic care. All participants will be required to complete a daily symptom diary until Day 14 and all participant will be asked to complete the Day 14 questionnaire, which will establish if any other members of the participant's household have developed symptoms of COVID-19. If a participant's symptoms clear before Day 14, they will be invited to complete the End of Illness questionnaire (healthcare use, adverse events, acceptability, infection in household contacts) on the day that these symptoms resolve, and continue to fill in the Daily Diary, in case of recurrence of symptoms until Day 14.

Participants who have been randomized to the Intervention arm, will be directed towards a password-protected webpage featuring videos and instructions on how to prepare the hypotonic saline solution and how to perform HSNIG, while those randomized to the Control arm will be directed towards a password-protected webpage featuring a video and instructions on how to perform ablution with plain water and gargling, as well as washing the nose other than ablution, but with plain (salt-free) clean water.

The patients who have been randomized to the intervention arm will be directed to the instructional video in which it will be explained that they should take 250 ml of clean water (water which has been boiled and cooled, or filtered or mineral water) in the measuring jug provided, and add one level teaspoon of salt (6.5 grams) and use this salty water for nasal washing and gargles. In order to standardize the study, and since sea-salt is not very commonly available in Pakistan, patients in the intervention arm will be provided sea salt (or preservative-free sodium chloride) for the treatment by the project, along with a measuring spoon calibrated at 6.5 grams of salt when filled level, and a graduated container showing 250 ml. This will be posted to them by courier as soon as they are randomized into the trial / intervention arm of the study. The addition of 6.5 grams of salt to 250 ml of water will make a 2.6% saline solution.

At consent, participants will be given the option to consent to the future collection of samples for COVID-19 serological analysis.

It is also proposed to randomly select approximately a proportion of all participants, according to availability of funds for testing for SARS-CoV-2 infection by RT-PCR, which will include a swab sample from the nose and/or the throat. to support the diagnosis of COVID-19. The selected participants will be informed of the government approved laboratories near their home which provide the required testing facilities and participants will be asked to pay the costs of these additional tests up front. The cost of the test and transport to the laboratory will be reimbursed to the participant after the participant sends the report of this test to the Allergy and Asthma Institute, Pakistan (AAIP), physically or electronically, and provides the original receipts of payment. Patients who have already had these tests done will be excluded from the random selection, and their results collected and recorded.

ELIGIBILITY:
INCLUSION CRITERIA

* Adults (≥18 years)
* Those living within larger cities of Pakistan (for laboratory access)
* Those self-isolating at home within 5 days of the start of the illness with:

  1. Clinical symptoms suggestive of COVID-19 (i.e. those who have at least one of the following symptoms: Respiratory symptoms, such as cough and shortness of breath; Fever; Muscle pain; Headache; Sore throat; New loss of taste or smell; Severe fatigue; Nausea or vomiting; Diarrhoea and Congestion or runny nose OR
  2. Those with virologically confirmed SARS-CoV-2 infection and clinical symptoms indicative of COVID-19 (as detailed in (a) above).
* Provision of informed consent

EXCLUSION CRITERIA

* Onset of illness (symptoms) more than 5 days
* Inability to consent
* Age less than 18 years.
* Pregnancy
* Immunosuppressed patients Inability to perform HSNIG
* Those taking part in another interventional medical trial
* Those with suspected/confirmed COVID-19 in whom hospital admission is recommended
* Those who do not have access to email / internet
* Those living in a household with another person currently participating in this study
* Those who have not provided consent to take part

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Time to resolution of symptoms | 2 weeks
  Self-reported time to resolution as assessed by completion of the validated self-reported UK-adapted short form of the Wisconsin Upper Respiratory Symptom Survey (WURSS-24) which will be used to collect daily symptom data

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Sheikh, MD, PhD, Study Chair — University of Edinburgh
Locations (1):
- The Allergy and Asthma Institute, Pakistan, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No
The study is anonymized, and individual participant data (IPD) will not be available to other researchers.

REFERENCES:
- [Derived] Yusuf OM, Ramalingam S, Norrie J, Graham C, Kakakhail A, Rextin AT, Baig RT, Yusuf SO, Ahmad B, Zahra S, Sheikh A. Hypertonic saline nasal irrigation and gargling for suspected or confirmed COVID-19: Pragmatic randomised controlled trial (ELVIS COVID-19). J Glob Health. 2024 Dec 13;14:05027. doi: 10.7189/jogh.14.05027. PMID 39666578